CLINICAL TRIAL: NCT05613816
Title: Prospective Data Collection to Compare Robotically Assisted Laparoscopy for Hysterectomies and Other Selected Indications in Comparison to Conventional Laparoscopy
Brief Title: Prospective Data Collection to Compare RAL for Hysterectomies and Other Indications in to Conventional Laparoscopy
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: MT_Asensus_Register
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Uterine Diseases
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Senhance Surgical System: 100 patients affected by uterine diseases with indication for hysterectomy undergo treatment with robotically assisted laparoscopic procedures using the Senhance Surgical System
  Interventions: Procedure: Senhance Surgical System

INTERVENTIONS:
Procedure: Senhance Surgical System — 100 patients affected by uterine diseases with indication for hysterectomy undergo treatment with robotically assisted laparoscopic procedures using the Senhance Surgical System

SUMMARY:
This is a prospective, single-center, observational clinical trial at the Department of Women's Health of the University Hospital Tübingen.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational clinical trial at the Department of Women's Health of the University Hospital Tübingen.

100 patients affected by uterine diseases with indication for hysterectomy undergo treatment with robotically assisted laparoscopic procedures using the Senhance Surgical System (See Synopsis - Indication A) and are compared to a cohort of 200 patients treated with conventional laparoscopic surgery from a similar ongoing study (Ethics vote: 621 /2018BO1).

100 patients affected by other uterine conditions / adnexal conditions that require uterine/adnexal/tubal surgery (see Synopsis - Indication B) undergo treatment with robotically assisted laparoscopic procedures using the Senhance Surgical System and are compared to a cohort of 200 patients with indication for other uterine conditions / adnexal conditions that require uterine/adnexal/tubal surgery (see Synopsis - Indication B) who underwent conventional laparoscopic surgery at the Department of Women's Health in the past.

At the end of patient recruitment, surgical procedure times, estimated blood loss, intra- and post-operative complications and the percentage of conversions from the robotic assisted treatment/conventional laparoscopic surgery to multiple access and/or to a laparotomic (open) approach will be documented.

Patients will answer questionnaires (German version of the Short Form-36health survey questionnaire (Medical Outcomes Trust), German version of the female sexual function index (FSFI)) at baseline and at 3 and 6 months of follow-up. A questionnaire for patient satisfaction will be answered one day post procedural, at discharge and at 3 and 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* BMI ≤40 kg/m2
* indication for hysterectomy for benign disease or prophylactic surgery due to hereditary cancer
* indication for radical hysterectomy and/or pelvic-/para-aortic (sentinel-node) lymphadenectomy for cervical cancer
* indication for modified radical hysterectomy and/or pelvic-/para-aortic (sentinel-node) lymphadenectomy for endometrial cancer
* indication for other uterine conditions / adnexal conditions that require uterine/adnexal/tubal surgery: Fibroids, Endometriomas, Cystic masses, Ectopic pregnancies, Sactosalpinx, Inflammatory adnexal disease, Opportunistic salpingectomy as part of hysterectomy or exclusively, Cervico-/Sacrokolpopexy
* size of uterus and vagina allows for retrieval by the vaginal route in cancer patients
* written informed consent

Exclusion Criteria:

* known extensive intra-abdominal adhesions
* anaesthesiological contraindications to laparoscopy
* women with pacemaker or other implants where electrosurgery is to be avoided
* women with known defects of the hemostasis
* pregnancy
* other internal or anatomical criteria that preclude a minimal invasive approach
* inability to understand patient information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
operating time | 60 minutes
  time from first incision to skin closure

SECONDARY OUTCOMES:
time under narcosis | 60 minutes
  duration of time in which the study participant is under the influence of a narcotic substance
console time | 60 minutes
  duration of time during which a surgeon is controlling the surgical robot from a console
estimated blood loss (milliliters) | 60 minutes
  using the following formula: ((Hemoglobin concentration preoperative (g/l)) - (Hemoglobin 1st day postoperative (g/l)))/((Hemoglobin preoperative (g/l)) - (Hemoglobin 1st day postoperative (g/l)))/2) × 1000
conversion to other surgical procedures (e. g. open) | 60 minutes
  if the original surgical plan during surgery is altered and switched to a different type of surgery to address unforeseen complications or difficulties that arise during the operation
time to discharge | 60 minutes
  length of time that a patient spends in the hospital before they are well enough to be released and sent home
intraoperative complications | 60 minutes
  (occurring during the surgical procedure)
perioperative complications | 24 hours
  (occurring less than 24h after the surgical procedure)
postoperative complications | 6 months
  (occurring more than 24h after the surgical procedure up to 6 months after surgical procedure)
German version of the Short Form-36health survey questionnaire (Medical Outcomes Trust) | at baseline, and at 3 and 6 months of follow-up
  The SF-36 questionnaire (Short Form 36 Health Survey) is a widely used measure of health status and quality of life. The questionnaire consists of 36 items that measure eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. The scores range from 0 to 100 for each domain, with higher scores indicating better health status. Therefore, higher scores on the SF-36 indicate a better outcome.
German version of the female sexual function index (FSFI) questionnaire | at baseline, and at 3 and 6 months of follow-up
  female sexual function index: a multidimensional self-report instrument for the assessment of female sexual function; The total composite sexual function score is a sum of domain scores and ranges from 2.0 (not sexually active and no desire) to 36.0. Higher scores on the FSFI indicate better sexual function.
Questionnaire for patient satisfaction | at one day post procedural, at discharge and at 3 and 6 months follow-up
  Including A Pain Score ( No Pain 0 - Worst Possible Pain 10) and B Satisfaction with: the severity of the pain; the quality of recovery; the scars; the surgery overall (Scale satisfaction: Extremely dissatisfied -- Dissatisfied -- Somewhat dissatisfied -- Neither satisfied nor dissatisfied -- Somewhat satisfied -- Satisfied -- Extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Andress, Dr, Principal Investigator — Department für Frauengesundheit am Universitätsklinikum Tübingen
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany